CLINICAL TRIAL: NCT06357637
Title: Preoperative Measurement of Abdominal Circumference as a Predictor of Difficult Spinal Anesthesia and Maternal Hypotension During Caesarian Section
Brief Title: Abdominal Circumference Measure in Caesarian Section
Acronym: ACirCuS
Status: Completed | Type: Observational
Sponsor: CHU Mohammed VI Marrakech (Other)
Responsible Party: Principal Investigator, Meryem Essafti, Assistant Professor, CHU Mohammed VI Marrakech
Other Study IDs: 59/2023
Record Dates: First submitted 2024-01-23; First posted 2024-04-10 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia, Spinal; Cesarean Section
Keywords: Preoperative evaluation; Abdominal circumference; Difficult spinal anesthesia; Maternal hypotension; Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measure of abdominal circumference — Measure of abdominal circumference preoperatively in both sitting and lying position

SUMMARY:
The goal of this observational study is to evaluate preoperative measures of abdominal circumference in patients admitted for a cesarean section. The main questions it aims to answer are:

* Can preoperative abdominal circumference predict patients with difficult spinal anesthesia
* Can preoperative abdominal circumference predict the occurrence of maternal hypotension during cesarean section Participants will be examined preoperatively in terms of visibility and palpation of spinous processes, abdominal circumference will be measured in the supine and sitting positions with other clinical parameters. Spinal anesthesia will be performed by the same experienced anesthesiologist with a standardized procedure. The number of skin punctures, needle reorientations, traumatic Cerebrospinal fluid, need for a paramedian approach or failure will be recorded. Maternal blood pressure and vasopressor requirements will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Parturients admitted for elective or emergency cesarean section

Exclusion Criteria:

* Acute fetal distress
* Umbilical cord prolapse
* Scoliosis
* Contraindication to spinal anesthesia
* Medical history of spinal surgery American Society of Anesthesia Status 4 or 5

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female pregnant patients
Study Population: Parturients scheduled for elective cesarean section or admitted for emergency cesarean section in the maternal operating theater of Mohammed VI University Hospital during the period of the study
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with difficult spinal anesthesia | During surgery
  More than two needle reorientations in the first puncture or more than one skin puncture

SECONDARY OUTCOMES:
Rate of Maternal hypotension | The first hour after spinal anesthesia is performed
  Systolic blood pressure below 90 mmHg or a drop of more than 20% of base value

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Mohammed VI, Marrakesh, Morocco

IPD SHARING:
Plan to Share IPD: Yes
All data collected throughout the trial will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 1 year after the publication of results
URL: https://www.chumarrakech.ma/

REFERENCES:
- [Background] Yu C, Gu J, Liao Z, Feng S. Prediction of spinal anesthesia-induced hypotension during elective cesarean section: a systematic review of prospective observational studies. Int J Obstet Anesth. 2021 Aug;47:103175. doi: 10.1016/j.ijoa.2021.103175. Epub 2021 May 1. PMID 34034957
- [Background] Merveille OC, Childers MK, Kreimid MM, George WD. Weaning from mechanical ventilation in a general rehabilitation center: a commentary. Am J Phys Med Rehabil. 1999 Jan-Feb;78(1):85-6. doi: 10.1097/00002060-199901000-00022. No abstract available. PMID 9923436

DOCUMENTS (2):
  • Study Protocol (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT06357637/Prot_000.pdf
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT06357637/ICF_001.pdf